CLINICAL TRIAL: NCT03955744
Title: Evaluation of 3D Translabial Ultrasound Imaging for Pessary Size Estimation
Brief Title: 3D Translabial Ultrasound for Pessary Size Estimation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor terminated study as there had been sufficient data collected from the recruited patients to characterize vaginal contraction biomechanics
Sponsor: Western University, Canada (Other)
Collaborators: Cosm Medical Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 113264; 6086 (Other: ReDA)
Record Dates: First submitted 2019-05-06; First posted 2019-05-20 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 3D translabial ultrasound (Experimental): 3D translabial ultrasound with concurrent vaginal manometry
  Interventions: Other: 3D translabial ultrasound

INTERVENTIONS:
Other: 3D translabial ultrasound — All patients will undergo 3D translabial ultrasound with vaginal manometry

SUMMARY:
This is a feasibility study looking at the use of 3D ultrasound with vaginal manometry at various distension volumes to predict the best available pessary for successful fit.

DETAILED DESCRIPTION:
Patients who are currently using a pessary for management of pelvic organ prolapse and who are able to remove/replace the pessary themselves will be approached for recruitment. The pessary will be removed two days prior to 3D translabial ultrasound. The vagina will be distended with a pressurized compliant bag with concurrent pressure and volume measurements. Translabial ultrasound will be used to measure structural parameters within the vagina at varying pressures/volumes. The volume, pressure and structural parameters measured will be compared to dimensions of the patient's own pessary to develop mathematical models to predict the best available pessary choice for the patient.

ELIGIBILITY:
Inclusion Criteria:

* are current pessary users (> 6 months) who have no pessary related complication, including discomfort, vaginal bleeding, and pessary extrusion
* are able to provide informed consent
* can perform self-care, i.e. removing and inserting the pessary themselves
* are willing to remove their pessary two days before the ultrasound examination date

Exclusion Criteria:

* inability to give informed consent
* inability to communicate with the person performing the consent and the sonographer performing ultrasound scanning
* history of pelvic radiation or surgery (excluding hysterectomy)
* using pessaries other than ring, incontinence dish, donut, Shaatz
* inability to perform the Valsalva maneuver or pelvic floor contraction
* restricted mobility that prevents them from ambulating to assess the comfort level of the pessary during the initial pessary fitting visit
* lack of sensation at the pelvic floor
* being pregnant at the time of the examination

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
3D ultrasound images and pressure/volume measurements of vagina in patients with pelvic organ prolapse | 1 hour and 20 minutes (i.e. the estimated time for the ultrasound and manometry examination per participant).
  3D ultrasound images of the vaginal canal and the pelvic floor will be obtained using various ultrasound probes. Pressure and volume measurements (i.e. manometry) will be obtained using a urodynamic system.

SECONDARY OUTCOMES:
Survey | 5 minutes
  Participants will be asked to fill out a short survey about their experience with the pessaries they already use and the ultrasound examination process

CONTACTS AND LOCATIONS:
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No